CLINICAL TRIAL: NCT05153291
Title: Electrically Guided Bachmann's Bundle Pacing Pilot Study: A Novel Lead Placement Strategy With Potential Antiarrhythmic Benefits
Brief Title: Electrically Guided Bachmann's Bundle Pacing: A Lead Placement Strategy With Potential Antiarrhythmic Benefits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Margaret Infeld, Cardiac Electrophysiology Fellow, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00001532
Record Dates: First submitted 2021-11-15; First posted 2021-12-10 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bachmann's bundle area pacing (Experimental): Lead placement in Bachmann's bundle area
  Interventions: Procedure: Bachmann's bundle lead placement
- Right atrial appendage pacing (Active Comparator): Lead placement in the right atrial appendage
  Interventions: Procedure: Right atrial appendage lead placement

INTERVENTIONS:
Procedure: Bachmann's bundle lead placement — Atrial lead placement at Bachmann's bundle area
  Arms: Bachmann's bundle area pacing
Procedure: Right atrial appendage lead placement — Atrial lead placement in the right atrial appendage
  Arms: Right atrial appendage pacing

SUMMARY:
Despite identification of optimal ventricular pacing sites, which not only avoid dyssynchronous activation but can restore ventricular synchrony, optimal atrial pacing sites have not yet been identified. Specialized conduction tracts do not exist in the atria as they do in the ventricle. Activating the atria in a manner that preserves or improves interatrial synchrony may provide clinical benefit based on recent data. Prior site-selective right atrial septal pacing (RAS) pacing studies relied on non-specific fluoroscopic guidance during lead placement. These studies were limited by the lack of an electrogram target and electrical measures of successful atrial resynchronization. The goal of this study is to prospectively evaluate Bachmann's bundle lead placement guided by fluoroscopy and electrical markers (an endocardial electrogram target and paced P-wave criteria) and determine its anti-arrhythmic efficacy compared with right atrial appendage (RAA) pacing. Patients presenting for pacemaker placement with an indication for an atrial lead are randomized to either electrically-guided BB lead placement or RAA lead placement and then followed for 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old
* Subject is referred for permanent pacemaker implantation with an indication for an atrial lead
* Subject has either paroxysmal atrial fibrillation or baseline intra-atrial conduction delay (P-wave duration >120ms on a 12-lead ECG)
* Subject is expected to remain available for standard-of-care pacemaker follow-up visits and study questionnaires

Exclusion Criteria:

* Subject has permanent atrial fibrillation or is in atrial fibrillation in the pre-operative area prior to the procedure (inability to assess paced P-wave morphology)
* Subject has pacemaker implantation prior to planned atrioventricular nodal ablation
* Subject has resting spontaneous sinus rate >85 beats-per-minute
* Subject has left ventricular ejection fraction <45%
* Subject is unable or unwilling to complete baseline or follow up quality of life questionnaires
* Subject is currently enrolled in a potentially confounding trial
* Subject is pregnant
* Subject's anticipated life expectancy is less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Atrial arrhythmia burden from pacemaker counters | Over 15 month follow up
  Derived from pacemaker counters and expressed as the average percentage of time per day in atrial fibrillation/tachycardia.

SECONDARY OUTCOMES:
Change in P-wave duration from sinus P-wave to paced P-wave in Bachmann's bundle and right atrial appendage lead groups | At implant
Atrial lead procedure time | At implant
Atrial lead fluoroscopy time | At implant
Atrial lead complications | Over 15 month follow up
Atrial lead capture threshold (Volts) | Over 15 month follow up
Atrial lead sensing threshold (millivolts) | Over 15 month follow up
Atrial lead impedance threshold (Ohms) | Over 15 month follow up
Atrial Fibrillation Severity Scale Version 2.0 | Over 15 month follow up
  Change in quality of life. The Atrial Fibrillation Severity Scale (AFSS) is composed of 19 items investigating four domains:
  1. AF burden (comprised of AF frequency + AF duration + AF severity): score range is 3-10, higher score = greater burden
  2. Health care utilization: score range is 0-7 for each question, higher score = more utilization
  3. Symptoms: score range is 0-35, higher score = greater symptom severity
  4. Global well-being: score range is 1-10, higher score = better quality of life
EQ-5D-3L survey (*EQ-5D-3L is the name of the instrument and is not an acronym) | Over 15 month follow up
  Change in quality of life. The EQ-5D-3L is a standardized instrument to assess generic health-related quality of life and contains questions on five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each of the five dimension, respondents are offered three response categories (no problems, some problems, extreme problems), leading to 243 possible health states. These health states are then converted into index based values (utilities) ranging from 0 to 1 by applying a valuation algorithm. The EQ-5D instrument includes a visual analogue scale (VAS), on which the patient is asked to score his/her current health state between 0 (worst imaginable health state) and 100 (best imaginable health state).
Hospitalization or urgent outpatient visit for atrial fibrillation | Within 15 months follow-up post pacemaker
Hospitalization or urgent outpatient visit for heart failure | Within 15 months follow-up post pacemaker
Cerebrovascular accident | Within 15 months follow-up post pacemaker
Atrial Fibrillation Ablation | Within 15 months follow-up post pacemaker
New start or up-titration of medications for the primary diagnosis of atrial fibrillation | Within 15 months follow-up post pacemaker

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data upon reasonable request